CLINICAL TRIAL: NCT00390338
Title: Phase I Evaluation of Alpha-Type-1 DC-Based and cDC-Based Intralymphatic Vaccines in Patients With Metastatic Melanoma
Brief Title: Vaccine Therapy in Treating Patients With Stage III or Stage IV Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pawel Kalinski (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Pawel Kalinski, Professor of Surgery and Immunology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-118; PCI-UPCI-03-118; NCI-7089; PCI-IRB-0409071; CDR0000504518 (Registry Identifier: PDQ (Physician Data Query)); NCI-2009-00125 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Melanoma (Skin)
Keywords: recurrent melanoma; stage IV melanoma; stage IIIA melanoma; stage IIIB melanoma; stage IIIC melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- peptide-pulsed type-1-polarized dendritic cells (Experimental): intralymphatic vaccination with peptide-pulsed type-1-polarized dendritic cells (aDC1)
  Interventions: Biological: polarized dendritic cells
- peptide-pulsed mature non-polarized dendritic cells (cDCs) (Experimental): intralymphatic vaccination with peptide-pulsed mature non-polarized dendritic cells (cDCs)
  Interventions: Biological: non-polarized dendritic cells

INTERVENTIONS:
Biological: polarized dendritic cells
  Arms: peptide-pulsed type-1-polarized dendritic cells
Biological: non-polarized dendritic cells
  Arms: peptide-pulsed mature non-polarized dendritic cells (cDCs)

SUMMARY:
RATIONALE: Vaccines made from a person's dendritic cells mixed with tumor peptides and proteins may help the body build an effective immune response to kill tumor cells. Infusing the vaccine directly into the lymphatic system may cause a stronger immune response and kill more tumor cells.

PURPOSE: This randomized phase I trial is studying the side effects and best dose of two dendritic cell vaccines in treating patients with stage III or stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the safety of intralymphatic autologous type-1-polarized dendritic cell vaccine vs autologous mature dendritic cell vaccine loaded with antigenic peptides and proteins in patients with stage III or IV melanoma.

Secondary

* Determine peripheral blood CD8+ and CD4+ T-cell responses to HLA-presented melanoma epitopes and autologous tumor cells using interferon gamma and interleukin-5 ELISPOT assay.
* Compare the delayed-type hypersensitivity (DTH) responses to these regimens and DTH to autologous tumor lysates in these patients.
* Compare the DTH response to keyhole limpet hemocyanin and pan-DR epitope (PADRE) in these patients.
* Correlate treatment-associated changes in immune response with clinical outcome.

OUTLINE: This is a randomized, open-label, dose-escalation study. Patients are randomized to 1 of 2 formulations of dendritic cell (DC) vaccines.

* Arm I: Patients receive intralymphatic autologous type-1-polarized (by interleukin-1-beta, tumor necrosis factor [TNF] alfa, interferon alfa, poly-I:C, and interferon gamma) DC vaccine that has been loaded with tumor-related peptide antigens (gp100:209-217[210M] peptide, tyrosinase peptide, MART-1:27-35 peptide, MAGE-3/6, and EphA2) and proteins (keyhole limpet hemocyanin [KLH; first course] or pan-DR epitope [PADRE] [second course]) every 6 hours on days 1-4 of weeks 1 and 6.
* Arm II: Patients receive intralymphatic autologous mature (by interleukin-1-beta, TNF alfa, interleukin-6, and prostaglandin E_2) DC vaccine that has been loaded with tumor-related peptide antigens and proteins as in arm I every 6 hours on days 1-4 of weeks 1 and 6.

Patients achieving complete response receive 2 more courses of treatment (3 months apart). Patients achieving partial response receive up to 10 more courses of treatment (1 month apart) in the absence of disease progression or unacceptable toxicity.

In each arm, cohorts of 4-7 patients receive escalating doses of DC vaccine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which no more than 1 of 7 patients experience dose-limiting toxicity.

Blood samples are obtained at baseline and periodically during and after treatment. Samples are examined by immunoenzyme techniques for immunologic measurements.

After completion of study therapy, patients are followed periodically for 10½ years and then annually thereafter.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathologically confirmed stage III or IVA (M1a) melanoma

  * Recurrent and inoperable disease
  * Any tumor thickness and any number of lymph nodes involved
  * Asymptomatic cutaneous and nodal disease allowed
  * Asymptomatic pulmonary metastatic disease (stage IVB, M1b) allowed
* No advanced symptomatic visceral disease, including any symptomatic visceral organ involvement, or disease associated with increased serum lactic dehydrogenase > 2.5 times upper limit of normal (stage IVC, M1c)
* Standard curative or palliative measures do not exist or are no longer effective
* Sufficient numbers of monocytes (≥ 20 x 10^6) must be obtained for the preparation of the vaccine

  * If an insufficient number of cells is obtained on first venipuncture, a second venipuncture may be performed (not exceeding 550 mL of blood within 8 weeks)
* No brain metastases by contrast-enhanced CT scan or MRI

  * Prior brain metastases allowed provided they were successfully treated and patient has been asymptomatic for ≥ 3 months
* HLA-A2 positive

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy ≥ 6 months
* Granulocyte count ≥ 1,500/mm³
* Lymphocyte count ≥ 500/mm³
* Platelet count > 70,000/mm³ (for venipuncture/pheresis procedure)
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN
* Gamma-glutamyl transferase ≤ 2.5 times ULN
* Lactic dehydrogenase ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* Bilirubin ≤ 1.5 times ULN
* No active infection
* No sensitivity to drugs that provide local anesthesia
* No pain uncontrolled by oral analgesics, including opiates and opiate analogs
* No active autoimmune disease
* No HIV, hepatitis B, or hepatitis C positivity
* Not pregnant or nursing
* Fertile patients must use effective contraception
* Negative pregnancy test
* No other malignancy except for nonmelanoma skin cancers or carcinoma in situ of the cervix, or other malignancy for which the patient has been continuously disease-free for ≥ 2 years

PRIOR CONCURRENT THERAPY:

* Recovered from prior surgery
* No radiotherapy, chemotherapy, or immunotherapy within the past 4 weeks (6 weeks for nitrosoureas or mitomycin C)
* No antibiotics within the past 7 days
* No systemic immunosuppressive agents, including steroids, within the past 4 weeks

  * Concurrent maintenance steroids for adrenal insufficiency allowed
* No other concurrent anticancer investigational or commercial agents or therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-10; Primary Completion 2012-05 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Safety of intralymphatic autologous type-1-polarized dendritic cell vaccine and autologous mature dendritic cell vaccine | 7 years

SECONDARY OUTCOMES:
Assess immune responses to each dendritic cell vaccine outcome | 7
  i. Peripheral blood CD8+ and CD4+ T cell responses against HLA-presented melanoma epitopes, and (in patients with available tumor tissue) against autologous tumor cells, and using IFNγ-, and IL-5- ELISPOT assays. CD8+ T cell responses (IFNγ ELISPOT) will be used as a secondary readout: the sum of the specific ELISPOT counts obtained (at week 8) with each of the individual HLA-A2-restricted peptides (less the respective counts obtained before the treatment), will be considered as a primary indication of the vaccine effectiveness.
  ii. Delayed type hypersensitivity (DTH) response to the mix of the melanoma-related peptides, injected intradermally in vivo, and DTH to autologous tumor lysates, in all cases when autologous tumor tissue is available.
  iii. Delayed type hypersensitivity (DTH) responses to KLH and PADRE injected intradermally in vivo.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad A. Tarhini, MD, MS, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - UPMC Cancer Center at Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania